CLINICAL TRIAL: NCT04703400
Title: Analysis of the Impact on Surgical Residency Programs in Times of Pandemic in Argentina: A Cross-sectional Study
Brief Title: Analysis of the Impact on Surgical Residency Programs in Times of Pandemic in Argentina
Status: Completed | Type: Observational
Sponsor: Clinica Universitaria Reina Fabiola, Universidad Catolica de Cordoba (Other)
Responsible Party: Principal Investigator, Palacios Huatuco, General Surgeon, Clinica Universitaria Reina Fabiola, Universidad Catolica de Cordoba
Other Study IDs: 0817040
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Surgical Education
Keywords: COVID-19; Surgical residents; Surgical training; Latin America
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: anonymous survey — anonymous survey with 25 mandatory questions

SUMMARY:
Introduction: COVID-19 emerged as a global pandemic in 2020 and affected teaching methods at all levels. Surgical education has also been significantly affected by this pandemic, but the effect remains unknown. We developed a survey with the aim of obtaining more information on how the COVID-19 pandemic affected the training and education of surgical residency programs in Argentina.

Material and methods: We carried out a cross-sectional study. We surveyed 195 resident physicians from various surgical residency programs, from August 15 to September 30, 2020, in Córdoba, Argentina. The effect of the COVID-19 pandemic on surgical training, academic program, and professional burnout of residents was analyzed.

DETAILED DESCRIPTION:
Introduction In 2020, the coronavirus disease (COVID-19) has affected more than 190 countries, registering more than 79.2 million cases and more than 1.7 million deaths worldwide since the start of the pandemic. The first reported case in Argentina was on March 5; two days later, the first fatality was registered in the country and in Latin America. On March 6, the first case of COVID-19 was confirmed in Córdoba, the second most populated province, out of a total of 23 provinces that make up the Argentine Republic. Until December 31, 2020, the Ministry of Health of the Province of Córdoba registered a total of 126,893 cases and 2,496 deaths from COVID-19.

The current health crisis produced by the coronavirus pandemic and defined as an unprecedented situation led us to raise doubts, controversies, and dilemmas in health care in general, and in surgery in particular, understanding that residents are possibly so vulnerable or more than all professionals.

In this scenario, the Association of Residents and Concurrents of General Surgery of Córdoba (ARCCC), which represents a non-profit civil association, founded in 1989, with the purpose of promoting scientific activity among resident physicians, prepared a survey with the objective of obtaining more information on how the COVID-19 pandemic affected the training and education of surgical residency programs in Córdoba.

Material and methods A cross-sectional study was carried out, supported by a digital survey tool (Google Forms). The survey presented 25 mandatory multiple-choice questions and was distributed through social networks such as WhatsApp, Facebook, and Instagram, from August 15 to September 30, 2020. All surgical residency programs in Córdoba, Argentina were invited to participate.

The survey asked the demographic characteristics of the residents, the type of hospital (public / private / Armed Forces) where they worked, the adherence of the training center to the resolution of the Ministry of Health 718/2020 (extension of discharge and promotion of the academic year of residents until September 30, 2020, within the health services, to attend the health and social emergency produced by COVID-19) (6), the type and the year (Considering the National Decree 718/2020) of the training program, work modality, number of days of attendance at your institution and surgical practices, before and during the pandemic. Residents were asked whether these changes would affect their surgical training and overall preparation for their next career move. The effects of the pandemic on the well-being and burnout of residents were also assessed.

All respondents voluntarily participated in this study and were advised that the information provided is confidential and will not be used to identify individual responses.

ELIGIBILITY:
Inclusion Criteria:

* medical residents
* both sexes (woman and man)
* residencies with surgical programs

Exclusion Criteria:

* residencies with medical clinic programs

Ages: 20 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: 195 respondents
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-01-03 (Actual)

PRIMARY OUTCOMES:
Demographic variables | August 15 to September 30, 2020
  gender and age
type of hospital | August 15 to September 30, 2020
  public / private / Armed Forces
type and year of training program | August 15 to September 30, 2020
  surgical program and position in residence
attendance at your institution and surgical practices | August 15 to September 30, 2020
  days and number of surgeries

CONTACTS AND LOCATIONS:
Locations (1):
- René M. Palacios Huatuco, Córdoba, Argentina

REFERENCES:
- [Background] Aziz H, James T, Remulla D, Sher L, Genyk Y, Sullivan ME, Sheikh MR. Effect of COVID-19 on Surgical Training Across the United States: A National Survey of General Surgery Residents. J Surg Educ. 2021 Mar-Apr;78(2):431-439. doi: 10.1016/j.jsurg.2020.07.037. Epub 2020 Jul 30. PMID 32798154
- [Background] Kogan M, Klein SE, Hannon CP, Nolte MT. Orthopaedic Education During the COVID-19 Pandemic. J Am Acad Orthop Surg. 2020 Jun 1;28(11):e456-e464. doi: 10.5435/JAAOS-D-20-00292. PMID 32282439
- [Background] Coe TM, Jogerst KM, Sell NM, Cassidy DJ, Eurboonyanun C, Gee D, Phitayakorn R, Petrusa E. Practical Techniques to Adapt Surgical Resident Education to the COVID-19 Era. Ann Surg. 2020 Aug;272(2):e139-e141. doi: 10.1097/SLA.0000000000003993. No abstract available. PMID 32675517
- [Background] Daodu O, Panda N, Lopushinsky S, Varghese TK Jr, Brindle M. COVID-19 - Considerations and Implications for Surgical Learners. Ann Surg. 2020 Jul;272(1):e22-e23. doi: 10.1097/SLA.0000000000003927. No abstract available. PMID 32345789
- [Background] Kim JY, Song JY, Yoon YK, Choi SH, Song YG, Kim SR, Son HJ, Jeong SY, Choi JH, Kim KM, Yoon HJ, Choi JY, Kim TH, Choi YH, Kim HB, Yoon JH, Lee J, Eom JS, Lee SO, Oh WS, Choi JH, Yoo JH, Kim WJ, Cheong HJ. Middle East Respiratory Syndrome Infection Control and Prevention Guideline for Healthcare Facilities. Infect Chemother. 2015 Dec;47(4):278-302. doi: 10.3947/ic.2015.47.4.278. Epub 2015 Dec 30. PMID 26788414
- [Background] Pelargos PE, Chakraborty A, Zhao YD, Smith ZA, Dunn IF, Bauer AM. An Evaluation of Neurosurgical Resident Education and Sentiment During the Coronavirus Disease 2019 Pandemic: A North American Survey. World Neurosurg. 2020 Aug;140:e381-e386. doi: 10.1016/j.wneu.2020.05.263. Epub 2020 Jun 5. PMID 32512244
- [Background] Kapila AK, Schettino M, Farid Y, Ortiz S, Hamdi M. The Impact of Coronavirus Disease 2019 on Plastic Surgery Training: The Resident Perspective. Plast Reconstr Surg Glob Open. 2020 Jul 1;8(7):e3054. doi: 10.1097/GOX.0000000000003054. eCollection 2020 Jul. PMID 32802694
- [Background] Huamanchumo-Suyon ME, Urrunaga-Pastor D, Ruiz-Perez PJ, Rodrigo-Gallardo PK, Toro-Huamanchumo CJ. Impact of the COVID-19 pandemic on general surgery residency program in Peru: A cross-sectional study. Ann Med Surg (Lond). 2020 Dec;60:130-134. doi: 10.1016/j.amsu.2020.10.031. Epub 2020 Oct 25. PMID 33133592
- [Background] Hewitt DB, Ellis RJ, Chung JW, Cheung EO, Moskowitz JT, Huang R, Merkow RP, Yang AD, Hu YY, Cohen ME, Ko CY, Hoyt DB, Bilimoria KY. Association of Surgical Resident Wellness With Medical Errors and Patient Outcomes. Ann Surg. 2021 Aug 1;274(2):396-402. doi: 10.1097/SLA.0000000000003909. PMID 32282379
- [Background] Bilimoria KY, Chung JW, Hedges LV, Dahlke AR, Love R, Cohen ME, Hoyt DB, Yang AD, Tarpley JL, Mellinger JD, Mahvi DM, Kelz RR, Ko CY, Odell DD, Stulberg JJ, Lewis FR. National Cluster-Randomized Trial of Duty-Hour Flexibility in Surgical Training. N Engl J Med. 2016 Feb 25;374(8):713-27. doi: 10.1056/NEJMoa1515724. Epub 2016 Feb 2. PMID 26836220